CLINICAL TRIAL: NCT00227539
Title: Early Positron Emission Tomography as a Predictor of Response in Neoadjuvant Chemotherapy for Non-Small Cell Lung Cancer
Brief Title: Positron Emission Tomography in Predicting Response in Patients Who Are Undergoing Treatment With Pemetrexed Disodium and Cisplatin With or Without Surgery for Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renato Martins, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6228; P30CA015704 (NIH); UWCC-6228; UWCC-UW-6228; UW-04033; LILY-UW-04033; CDR0000441239 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed; Chemotherapy, Adjuvant; Fluorodeoxyglucose F18

ARMS (1):
- Neoadjuvant therapy, PET scan and surgery (Experimental)
  Interventions: Drug: cisplatin; Drug: pemetrexed disodium; Procedure: adjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Drug: cisplatin
Drug: pemetrexed disodium
Procedure: adjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET), (done before, during, and after chemotherapy) may help doctors predict a patient's response to treatment and help plan the best treatment. Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well PET works in predicting response in patients who are undergoing treatment with pemetrexed disodium and cisplatin with or without surgery for stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of fludeoxyglucose F 18 positron emission tomography in predicting radiological and pathological response in patients treated with pemetrexed disodium and cisplatin with or without surgery for stage IB-IIIB non-small cell lung cancer (NSCLC).

Secondary

* Determine the safety of cisplatin and pemetrexed disodium in these patients.
* Determine the radiographic response rate, duration of response, and time to progression in patients treated with cisplatin and pemetrexed disodium.

OUTLINE: This is a multicenter study.

* Fludeoxyglucose F 18 (18FDG) positron emission tomography (PET) imaging: All patients undergo positron emission tomography (PET) imaging of the head, neck, thorax, abdomen, and pelvis. Patients receive fludeoxyglucose F 18 (^18FDG) IV followed by 45 minutes of rest. PET imaging is done over 1 hour and 8 minutes. Patients undergo PET imaging at three points during the study: 4 weeks prior to treatment, after the first cycle of treatment, and after 3 courses of chemotherapy. Some patients then undergo surgical resection of the tumor.
* Chemotherapy: Patients receive cisplatin IV over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Stage IB, II, IIIA, or IIIB (T4, N0-1) disease

  * Staging must have been performed 4 weeks prior to study entry with a CT scan of chest, upper abdomen, and fludeoxyglucose F 18 (^18FDG) positron emission tomography (PET) scan
  * Mediastinal evaluation and staging based on combination of CT scan and FDG-PET results
* If N1 or N2 nodes are found by FDG-PET or CT scan, metastases must be ruled out by brain MRI
* Measurable and resectable disease

  * T4 lesions must be resectable
* Eligible for curative surgery
* No malignant pleural effusion

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,250/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3.0 times ULN

Renal

* Creatinine clearance ≥ 45 mL/min

Pulmonary

* Adequate pulmonary reserve to undergo surgery

  * Predicted FEV_1 > 0.8 L after resection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to take corticosteroids
* Able to take folic acid or vitamin B_12 supplements
* No other malignancy within the past 5 years except nonmelanoma skin cancer or noninvasive cervical cancer
* No concurrent serious or uncontrolled disorder that would preclude study participation
* No type I diabetes mellitus

  * Type II diabetes mellitus allowed if glucose is 80-150 mg/dL

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent thrombopoiesis-stimulating agents

Chemotherapy

* At least 5 years since prior chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy

Radiotherapy

* No prior radiotherapy to the chest
* No concurrent curative or palliative radiotherapy

Surgery

* Not specified

Other

* At least 30 days since prior non-FDA-approved or investigational agents
* At least 5 days since prior aspirin or other nonsteroidal anti-inflammatory agents (8 days for long-acting agents [e.g., piroxicam])
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-07; Primary Completion 2010-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, MD, MPH, Principal Investigator — Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Derived] Romine PE, Martins RG, Eaton KD, Wood DE, Behnia F, Goulart BHL, Mulligan MS, Wallace SG, Kell E, Bauman JE, Patel SA, Vesselle HJ. Long term follow-up of neoadjuvant chemotherapy for non-small cell lung cancer (NSCLC) investigating early positron emission tomography (PET) scan as a predictor of outcome. BMC Cancer. 2019 Jan 14;19(1):70. doi: 10.1186/s12885-019-5284-2. PMID 30642285

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Therapy, PET Scan and Surgery: cisplatin
  pemetrexed disodium
  adjuvant therapy
  therapeutic conventional surgery
  fludeoxyglucose F 18
Period: Overall Study
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Started | 25
Completed | 24
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Positron Emission Tomography as a Predictor of Response Measured by the Decrease in Standard Uptake Variable (SUV) After 1 Course of Therapy
Description: Number of Participants with Decrease in Standard Uptake Variable (SUV) After 1 Course of Therapy
Time Frame: Between days 18 and 22 prior to second chemotherapy infusion
Population: Only 19 patients had PET scans at both baseline and day 18-22 available for review.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Number analyzed (Participants) | 19
Participants | 11

2. Secondary Outcome: Safety of Neoadjuvant Chemotherapy
Description: The number of patients that experienced a grade 3 or higher adverse event.
Time Frame: Up to 4 weeks after last dose of chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Number analyzed (Participants) | 25
Participants | 10

3. Secondary Outcome: Efficacy of Neoadjuvant Chemotherapy as Measured by Radiologic Response Rate
Description: The number of patients that had either a CR, PR or SD after the completion of chemotherapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Up to 4 weeks after last dose of chemotherapy
Population: One patient was excluded from the efficacy analysis because they were subsequently found to be ineligible. Three patients were unevaluable because they did not have have a CT scan after the completion of chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Number analyzed (Participants) | 21
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first dose of chemotherapy through 4 weeks following the final dose of chemotherapy.
Description: Only grade 3 and higher adverse events were collected.
Arm/Group | Neoadjuvant Therapy, PET Scan and Surgery
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Therapy, PET Scan and Surgery (N=25)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Therapy, PET Scan and Surgery (N=25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (25)
Fatigue (General disorders) | 7 (25)
Drug Reaction (Immune system disorders) | 3 (25)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (25)
Pain (Nervous system disorders) | 2 (25)
Nausea (Gastrointestinal disorders) | 2 (25)
pneumonia (Infections and infestations) | 1 (25)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (25)
Vomiting (Gastrointestinal disorders) | 1 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes